CLINICAL TRIAL: NCT03573310
Title: A Phase 1, First-in-Human, Open-Label Study of the Safety, Pharmacokinetics, and Pharmacodynamics of JNJ-64619178, an Inhibitor of Protein Arginine Methyltransferase 5 (PRMT5) in Subjects With Advanced Cancers
Brief Title: A Study of JNJ-64619178, an Inhibitor of PRMT5 in Participants With Advanced Solid Tumors, NHL, and Lower Risk MDS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR108485; 64619178EDI1001 (Other: Janssen Research & Development, LLC); 2018-000067-87 (EudraCT Number); 2024-515254-24-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2018-06-20; First posted 2018-06-29 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Neoplasms; Solid Tumor, Adult; Non-Hodgkin Lymphoma; Myelodysplastic Syndromes
Keywords: Lower risk MDS; Low risk MDS; Lower-risk MDS; Low-risk MDS; Intermediate 1 risk MDS; Intermediate-1 risk MDS
MeSH Terms: conditions — Neoplasms; Lymphoma, Non-Hodgkin; Myelodysplastic Syndromes | interventions — JNJ-64619178

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose escalation and RP2D Selection (Experimental): Participants with solid tumors or non-Hodgkin lymphoma (NHL) will receive JNJ-64619178 orally as per the assigned sequential cohorts and doses will be escalated based on the review of all available data including, but not limited to, pharmacokinetic, pharmacodynamic, safety, and clinical activity. One or more recommended Phase 2 dose(s) (RP2Ds) may be determined for further exploration.
  Interventions: Drug: JNJ-64619178
- Part 2:Dose Confirmation and Expansion (Experimental): Participants with myelodysplastic syndromes (MDS) will receive JNJ-64619178 at a dose less than or equal to the RP2D selected in Part 1 for 24 weeks, or longer if there is evidence of clinical benefit. The dose level of JNJ-64619178 may be adjusted based on observed toxicities.
  Interventions: Drug: JNJ-64619178

INTERVENTIONS:
Drug: JNJ-64619178 — JNJ-64619178 capsules to be administered orally.

SUMMARY:
The purpose of the study is to identify the maximum tolerated dose (MTD) of JNJ-64619178 in participants with relapsed/refractory B cell non-Hodgkin lymphoma (NHL) or advanced solid tumors and also to identify the recommended Phase 2 dose(s) (RP2Ds) of JNJ-64619178 for NHL and advanced solid tumors (Part 1) and to confirm the tolerability of JNJ-64619178 in participants with lower risk myelodysplastic syndromes (MDS) (Part 2).

DETAILED DESCRIPTION:
The study is designed to determine the maximum tolerated dose (MTD) of JNJ-64619178, and to select a dose(s) and regimen(s) that may be used in future clinical development. Study evaluations will include safety, pharmacokinetics, biomarkers and efficacy evaluations (Disease Assessments). Adverse events will be evaluated throughout the study. The study is divided into 4 periods: a screening phase, a pharmacokinetic run-in phase, a treatment phase, and a post treatment follow-up phase. An end-of-treatment visit will be completed less than or equal (<=) 30 days (+7 days) after the last dose of study drug or prior to the start of a new anticancer therapy, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* B cell non-Hodgkin lymphoma (NHL) or solid tumors, or lower risk MDS
* At least 1 measurable site of disease for B cell-NHL and solid tumors
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* Adequate organ function
* Women of childbearing potential must have a negative highly sensitive serum (beta-human chorionic gonadotropin [beta-hCG]) at screening and prior to the first dose of study drug. Women must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for a period of 90 days after receiving the last dose of study drug

Exclusion Criteria:

* History of, or known, central nervous system (CNS) involvement
* Prior solid organ transplantation
* Either of the following: a) Received an autologous stem cell transplant less than or equal (<=) 9 months before the first dose of study drug B) Prior treatment with allogenic stem cell transplant
* History of malignancy (other than the disease under study) within 3 years before the first administration of study drug. Exceptions include squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy that in the opinion of the investigator, with concurrence with the sponsor's medical monitor, is considered cured with minimal risk of recurrence within 3 years
* Known allergies, hypersensitivity, or intolerance to JNJ-64619178 or its excipient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2025-09-25 (Actual); Study Completion 2025-09-25 (Actual)

PRIMARY OUTCOMES:
Part 1 and Part 2: Number of Participants with Dose-limiting Toxicities (DLTs) | Approximately 3 years
  DLTs are defined as certain non-hematologic and hematologic toxicities of Grade 3 or higher.

SECONDARY OUTCOMES:
Part 1 and Part 2: Number of Participants with Adverse Events (AE) | Approximately 3 years
  AE is any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship.
Part 1 and Part 2: Number of Participants with AE by Severity | Approximately 3 years
  Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE). Severity scale ranges from Grade 1 (Mild) to Grade 4 (Life-threatening). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event.
Part 1 and Part 2: Number of Participants with Abnormal Vital Signs | Approximately 3 years
  Number of participants with abnormality in vital signs (temperature, pulse/heart rate, and blood pressure) will be reported.
Part 1 and Part 2: Number of Participants with Laboratory Abnormalities | Approximately 3 years
  Number of participants with laboratory abnormalities (serum chemistry, hematology, and coagulation, and disease-related laboratory abnormalities) will be reported.
Part 1 and Part 2: Number of Participants with Electrocardiogram (ECG) Abnormalities | Approximately 3 years
  Number of participants with electrocardiogram(ECG) abnormalities will be reported.
Part 1 and Part 2: Maximum Plasma Concentration (Cmax) of JNJ-64619178 | Approximately 3 years
  Cmax is the maximum observed plasma concentration.
Part 1 and Part 2: Area Under the Plasma Concentration Versus Time Curve From Time Zero to End of Dosing Interval (AUCtau) | Approximately 3 years
  AUCtau is the measure of the plasma drug concentration from time zero to end of dosing interval.
Part 1 and Part 2: Minimum Plasma Concentration (Cmin) | Approximately 3 years
  Cmin is the minimum observed plasma concentration.
Part 1 and Part 2: Plasma Decay Half-Life (t1/2) | Approximately 3 years
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Part 1 and Part 2: Volume of Distribution at Steady-State Influenced by the Fraction Absorbed (Vss/F) | Approximately 3 years
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Steady state volume of distribution (Vss) is the apparent volume of distribution at steady state which is estimated by (D/AUC[0-infinity])* (AUMC[0-infinity])/(AUC[0-infinity]) where D is the dose of study drug, AUMC(0-infinity) is the area under the first moment curve extrapolated to infinity and AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time. All these parameters will be assessed as influenced by the fraction absorbed.
Part 1 and Part 2: Apparent Total Systemic Clearance of Drug (CL/F) after Extravascular Administration | Approximately 3 years
  Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Part 1 and Part 2: Accumulation Index (RA) | Approximately 3 years
  Accumulation Index (RA) is calculated as AUC (0-24) value at steady state divided by AUC (0-24) value after first dose.
Part 1 and Part 2: Plasma Concentration of Symmetric Dimethyl-Arginine (SDMA) | Approximately 3 years
  Plasma concentration of symmetric dimethyl-arginine (SDMA) will be evaluated.
Part 1: Percentage of Participants with B cell non-Hodgkin lymphoma (NHL) Showing Overall Response of Partial Response (PR) or Better | Approximately 3 years
  Overall response rate (ORR) is defined as the percentage of participants who have a PR or better. Per Lugano classification, PR is defined as greater than or equal (>=) 50 percent (%) decrease in size of target lesions.
Part 1: Percentage of Participants with Solid Tumors Showing Overall Response of PR or Better | Approximately 3 years
  Overall response rate (ORR) is defined as the percentage of participants who have a PR or better. PR criteria in solid tumors (RECIST) is >= 30 percent (%) decrease in the sum of the diameters of all index lesions compared with baseline in 2 observations at least 4 weeks apart, in absence of new lesions or unequivocal progression of non-index lesions.
Part 1: Duration of Response | Approximately 3 years
  Duration of response (DOR) will be calculated from the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease (PD), as defined in the disease-specific response criteria, or death due to any cause, whichever occurs first. PD (per RECIST 1.1) defined as at least 20% increase in the sum of the longest diameters of index lesions or unequivocal progression of non-index lesions. Per Lugano classification, PD: target lesions larger; clear progression of non-target lesions; or new tumor lesions; new or recurrent bone marrow involvement; splenomegaly + 2 centimeter (cm) or +50%.
Part 1: Clinical Benefit Rate | Approximately 3 years
  Clinical benefit rate is defined as percentage of participants who have a complete response (CR), PR and sustained stable disease of 12 weeks or more. Sustained stable disease of 12 weeks or more is defined as participants with stable disease assessment maintained for about 12 weeks or longer from baseline. Per Lugano classification CR is defined as no detectable disease by computed tomography (CT) or positron emission tomography (PET)/CT scan. Evaluation criteria as per RECIST 1.1 for CR is defined as disappearance of all lesions in 2 consecutive observations not less than 4 weeks apart.
Part 2: Red Blood Cell (RBC) Transfusion Independence (TI) Rate | Approximately 3 years
  Percentage of participants with TI, defined as being without any transfusion during any consecutive 8 weeks (56 days) between the first dose of study drug and treatment discontinuation.
Part 2: Overall Improvement Rate | Approximately 3 years
  Overall improvement rate is defined as the percentage of participants achieving complete remission (bone marrow: less than or equal to (<=)5% myeloblasts with normal maturation of all cell lines; Peripheral blood: hemoglobin >=11 gram per deciliter (g/dL); platelets >=100*109/liter(L); neutrophils >=1.0*109/L; blasts, 0%), partial remission (All complete remission criteria if abnormal before treatment except: Bone marrow blasts decreased by >=50% over pretreatment but still >5% Cellularity and morphology not relevant), or hematologic improvement (HI) (Erythroid response [pretreatment, <11 g/dL]; Platelet response (pretreatment, <100*10^9/L); Neutrophil response (pretreatment, <1*10^9/L); Progression or relapse after HI) according to modified International Working Group (IWG) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (18):
- United States (4):
  - Florida Specialist and Cancer Institute, Sarasota, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Ohio State University, Columbus, Ohio
  - University of Texas, MD Anderson Cancer Center, Houston, Texas
- Canada (2):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Princess Margaret Cancer Centre University Health Network, Toronto, Ontario
- Germany (3):
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Goethe Universität Frankfurt, Frankfurt am Main
  - Universitaetsklinikum Leipzig, Leipzig
- Israel (3):
  - Carmel Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Tel Aviv Sourasky MC, Tel Aviv
- Spain (6):
  - Hosp. Univ. Germans Trias I Pujol, Badalona
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Clinica Univ. de Navarra, Pamplona
  - Hosp Clinico Univ de Salamanca, Salamanca
  - Hosp. Virgen Del Rocio, Seville